CLINICAL TRIAL: NCT00180895
Title: A Phase II Study of Mabthera (Rituximab) in Children and Adolescents With Relapsed and Refractory B-Cell NHL/L3ALL
Brief Title: Rituximab in Children and Adolescents With Relapsed and Refractory B-Cell NHL/L3ALL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rituximab childhood
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Burkitt Lymphoma
Keywords: Burkitt lymphoma; B-cell non Hodgkin lymphoma; B-cell ALL; Refractory; Relapse; Rituximab; Children
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, B-Cell; Recurrence | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
This is a multicentric phase II study of Mabthera (rituximab) in children and adolescents with relapsed and refractory B-cell NHL/L3ALL. The primary objective is to determine the response rate of Rituximab as single agent in relapsed or refractory Burkitt lymphoma, L3 acute leukemia, large B-cell lymphoma and non subclassified aggressive B-cell NHL

DETAILED DESCRIPTION:
This is a multicentric phase II study of Mabthera (rituximab) in children and adolescents with relapsed and refractory B-cell NHL/L3ALL. The primary objective is to determine the response rate of Rituximab as single agent in relapsed or refractory Burkitt lymphoma, L3 acute leukemia, diffuse large B-cell lymphoma and non subclassified aggressive B-cell NHL. The secondary objectives are to assess the toxicity profile of Rituximab in children and adolescents as single agent, and when followed by chemotherapy, to study pharmacokinetics of Rituximab in serum and in CSF and to determine the overall duration of response, time to progression and survival in patients responders to antiCD20 initially alone and followed by chemotherapy.

Patients will receive Rituximab (Mabthera) at 375 mg/m2, once a week during 4 weeks, administered in IV infusion starting at 50mg/h and increasing by steps of 50 mg/h every 30mn until the speed of 400 mg/h. Patients with combined CNS relapse will receive an intrathecal injection of MTX+HC+Ara-C 48 h after each injection of rituximab First assessment will be done prior to receiving the 3rd course of rituximab. Responding patients (CR, PR) and patients with objective effect (OE) will receive the 3rd and 4th injections of rituximab before starting the salvage chemotherapy (COPADM, CYVE/CC course or ICE, depending on previous chemotherapy regimen received by the patient, followed by HDCT+ hematopoietic stem cell rescue). A second evaluation will be done after the 4th course if performed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven B-cell malignancies, either Burkitt NHL or L3 ALL or large B-cell lymphoma or aggressive B-cell NHL, with the exception of diffuse large B-cell lymphoma arising in the mediastinum.
* Immunohistochemistry showing CD20 positivity
* Measurable (at least one bi-dimensionally measurable lesion) or evaluable (bone marrow, bone involvement) disease in progression since the last evaluation
* First relapsed or refractory disease after LMB or BFM protocol, except the isolated CNS relapses
* Life expectancy > 4 weeks
* Performance status (Karnofsky) > 30
* Adequate hepatic, renal and cardiac functions
* Wash out of 3 weeks in case of recent chemotherapy
* Complete initial work-up within 8 days prior to treatment
* Able to comply with scheduled follow-up and with management of toxicity
* Written inform consent form from adult patients and from parents and legal guardians for minor children

Exclusion Criteria:

* Active viral infection, especially chronic hepatitis B
* previous salvage therapy for relapse
* Prior or current history of severe allergy
* Primary large B-cell lymphoma of the mediastinum
* Isolated CNS relapse

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2004-06

PRIMARY OUTCOMES:
Rate of patients achieving at least objective response after 2 courses of rituximab

SECONDARY OUTCOMES:
Rate of objective response after 4 courses of rituximab
Rate of initially responding patients who progressed during the second phase of treatment
Toxicity
Pharmacokinetic evaluation in serum and CSF

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Patte, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France